CLINICAL TRIAL: NCT03638167
Title: Phase 1 Study of EGFR806-specific CAR T Cell Locoregional Immunotherapy for EGFR-positive Recurrent or Refractory Pediatric Central Nervous System Tumors
Brief Title: EGFR806-specific CAR T Cell Locoregional Immunotherapy for EGFR-positive Recurrent or Refractory Pediatric CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrainChild-02
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Tumor, Pediatric; Glioma; Ependymoma; Medulloblastoma; Germ Cell Tumor; Atypical Teratoid/Rhabdoid Tumor; Primitive Neuroectodermal Tumor; Choroid Plexus Carcinoma; Pineoblastoma
Keywords: CNS, CAR T cell, EGFR-positive; pediatric, young adults, brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Ependymoma; Medulloblastoma; Neoplasms, Germ Cell and Embryonal; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Choroid Plexus Carcinoma; Pinealoma; Brain Neoplasms | interventions — Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM A (Tumor Cavity Infusion) (Experimental): Patients with supratentorial tumors for which CAR T cells will be delivered into the tumor resection cavity
  Interventions: Biological: EGFR806-specific chimeric antigen receptor (CAR) T cell
- ARM B (Ventricular System Infusion) (Experimental): Patients with either infratentorial tumors or leptomeningeal tumors for which the CAR T cells will be delivered into the fourth ventricle or lateral ventricle, respectively
  Interventions: Biological: EGFR806-specific chimeric antigen receptor (CAR) T cell

INTERVENTIONS:
Biological: EGFR806-specific chimeric antigen receptor (CAR) T cell — Autologous CD4+ and CD8+ T cells lentivirally transduced to express an EGFR806 specific chimeric antigen receptor (CAR) and EGFRt given via indwelling central nervous system (CNS) catheter

SUMMARY:
This is a Phase 1 study of central nervous system (CNS) locoregional adoptive therapy with autologous CD4+ and CD8+ T cells that are lentivirally transduced to express an EGFR806 specific chimeric antigen receptor (CAR) and EGFRt. CAR T cells are delivered via an indwelling catheter into the tumor cavity or the ventricular system in children and young adults with recurrent or refractory EGFR-positive CNS tumors. The primary objectives of this protocol are to evaluate the feasibility, safety, and tolerability of CNS-delivered fractionated CAR T cell infusions employing intra-patient dose escalation. Subjects with supratentorial tumors will receive sequential EGFR806-specific CAR T cells delivered into the tumor resection cavity, subjects with infratentorial tumors will receive sequential CAR T cells delivered into the fourth ventricle, and subjects with leptomeningeal disease will receive sequential CAR T cells delivered into the lateral ventricle. The secondary objectives are to assess CAR T cell distribution within the cerebrospinal fluid (CSF), the extent to which CAR T cells egress into the peripheral circulation, and EGFR expression at recurrence of initially EGFR-positive tumors. Additionally, tumor response will be evaluated by magnetic resonance imaging (MRI) and CSF cytology. The exploratory objectives are to analyze CSF specimens for biomarkers of anti-tumor CAR T cell presence and functional activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 15 and ≤ 26 years
2. Histologically diagnosed EGFR positive Central Nervous System (CNS) tumor
3. Evidence of refractory or recurrent CNS disease for which there is no standard therapy
4. Able to tolerate apheresis or apheresis product available for use in manufacturing
5. CNS reservoir catheter, such as an Ommaya or Rickham catheter
6. Life expectancy ≥ 8 weeks
7. Lansky or Karnofsky score ≥ 60
8. If patient does not have previously obtained apheresis product, patient must have recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy and discontinue the following prior to enrollment:

   1. ≥ 7 days post last chemotherapy/biologic therapy administration
   2. 3 half lives or 30 days, whichever is shorter post last dose of anti-tumor antibody therapy
   3. Must be at least 30 days from most recent cellular infusion
   4. All systemically administered corticosteroid treatment therapy must be stable or decreasing within 1 week prior to enrollment with maximum dexamethasone dose of 2.5 mg/m2/day. Corticosteroid physiologic replacement therapy is allowed.
9. Adequate organ function
10. Adequate laboratory values
11. Subjects of childbearing/fathering potential must agree to use highly effective contraception

Exclusion Criteria:

1. Diagnosis of classic diffuse intrinsic pontine glioma (DIPG)
2. Presence of ≥ Grade 3 cardiac dysfunction or symptomatic arrhythmia requiring intervention
3. Presence of primary immunodeficiency/bone marrow failure syndrome
4. Presence of clinical and/or radiographic evidence of impending herniation
5. Presence of active malignancy other than the primary CNS tumor under study
6. Presence of active severe infection
7. Receiving any anti-cancer agents or chemotherapy
8. Pregnant or breastfeeding
9. Subject and/or authorized legal representative unwilling to provide consent/assent for participation in the 15 year follow up period
10. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Safety: any adverse events associated with one or multiple EGFR806-specific CAR T cell product infusions will be assessed by CTCAE v5.0. | up to 6 months
  The type, frequency, severity, and duration of adverse events as a result of EGFR806-specific CAR T cell infusion will be summarized
Feasibility: The number of successfully manufactured and infused EGFR806-specific CAR T cell product | 28 days
  The proportion of products successfully manufactured and infused will be measured

SECONDARY OUTCOMES:
CAR T cell distribution: The number of subjects with CAR T cell persistence in the cerebrospinal fluid (CSF) and peripheral blood as measured by flow cytometry | up to 6 months
  The trafficking of the EGFR806-specific CAR T cell product through the CSF by measuring remaining CAR T cells from a prior infusion at the time of each infusion and the trafficking of EGFR806-specific CAR T cells from the CSF into the peripheral blood will be evaluated.
Expression of target epitope: assessment of whether EGFR expression changes in relapsed CNS tumors that were EGFR positive prior to treatment with CAR T cells via immunohistochemistry on resected tissue samples. | 28 days
  The changes in EGFR expression at diagnosis and recurrence of central nervous system (CNS) tumors, if samples from multiple time points is available, will be investigated by evaluating pathology specimens from previous surgeries
Disease response: Assessment of disease response of EGFR-expressing refractory or recurrent central nervous system (CNS) tumors to EGFR806 specific CAR T cell therapy delivered directly into the CNS by cytology and radiology criteria. | up to 6 months
  The response of recurrent or refractory central EGFR-expressing CNS tumors to EGFR806-specific CAR T cell therapy delivered directly into the CNS will be determined by evaluating CSF for tumor cells and by CNS imaging with MRIs.

OTHER OUTCOMES:
Quantitative biomarker assessment of anti tumor CAR T cell functional activity | up to 6 months
  The presence of biomarkers of anti-tumor CAR T cell functional activity, such as cytokines, will be quantified via protein expression analysis in CSF. These findings will be correlated with safety determined by the occurrence of adverse events, and response by disease evaluations via CSF cytology and MRI imaging of the CNS.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Gust, MD, PhD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No